CLINICAL TRIAL: NCT05577273
Title: Does Antibiotic Prophylaxis at Urinary Catheter Removal Prevent Urinary Tract Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Omri Schwarztuch Gildor (Other)
Responsible Party: Sponsor-Investigator, Omri Schwarztuch Gildor, Principal Investigator, Clalit Health Services
Organization: Clalit Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MMC-0048-18
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Urologic Diseases; Urinary Tract Disease
MeSH Terms: conditions — Urologic Diseases | interventions — cefuroxime axetil; Trimethoprim

STUDY DESIGN:
Intervention Model Description: 2 arms: antibiotic prophylaxis vs no treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic prophylaxis (Experimental): Single dose of p.o. antibiotic given 1 hour before catheter removal. The antibiotic of choice is Cefuroxime axetil 500 mg. For penicillin allergy, trimethoprim/sulfamethoxazole 160mg/800mg.
  Interventions: Drug: Cefuroxime axetil (trimethoprim/sulfamethoxazole if penicillin allergy)
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Cefuroxime axetil (trimethoprim/sulfamethoxazole if penicillin allergy) — single dose of P.O. Cefuroxime Axetil 500 mg. For penicillin allergy patients, single dose of P.O. Trimethoprim/Sulfamethoxazole 160mg/800mg
  Arms: Antibiotic prophylaxis

SUMMARY:
At the end of most urological procedures, the doctor inserts a urethral catheter for a period of up to 5 days. According to AUA's guidelines, prophylactic antibiotic is indicated during catheter removal.

The aim of our study is to check the influence of the antibiotic treatment on urinary tract infections after catheter removal

ELIGIBILITY:
Inclusion Criteria:

* performing urological operation for other reason

Exclusion Criteria:

* cannot give informed consent
* <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
UTI | 30 day
  Number of participants with primary care/emergency department visits because of dysuria, fever, chills or other UTI related symptoms

SECONDARY OUTCOMES:
positive culture approved UTI | 30 day
  Number of participants with primary care/emergency department visits because of dysuria, fever, chills or other UTI related symptoms, and a positive urine/blood culture taken during the time frame
Hospitalizations due to UTI | 30 day
Bacteremia | 30 day
  Number of patients admitted to the hospital, that have at least 1 positive blood culture

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No